CLINICAL TRIAL: NCT00005033
Title: Phase II Study of Recombinant Humanized Monoclonal Antibody Against HER2 for the Treatment of Recurrent Osteosarcoma
Brief Title: Trastuzumab in Treating Patients With Recurrent Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067558; MSKCC-99097; NCI-T98-0083
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2004-08

CONDITIONS: Sarcoma
Keywords: recurrent osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Trastuzumab

INTERVENTIONS:
Biological: trastuzumab
Procedure: conventional surgery

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of trastuzumab in treating patients who have recurrent osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, freedom from progression, and survival of patients with recurrent osteosarcoma when treated with trastuzumab (Herceptin).
* Evaluate the toxicity of this drug in young patients with a history of osteosarcoma and prior therapy with doxorubicin.

OUTLINE: This is a multicenter study.

Patients receive trastuzumab (Herceptin) IV over 30-90 minutes weekly. Treatment continues for up to 52 weeks in the absence of disease progression or unacceptable toxicity. After approximately 12 weeks of treatment, patients are evaluated for response and undergo surgical resection if clinically appropriate.

Patients are followed for 1 year for survival.

PROJECTED ACCRUAL: Approximately 20-40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent osteosarcoma after initial systemic therapy with doxorubicin
* Measurable disease
* Immunohistochemical evidence of 2+ overexpression of HER2

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* ALT or AST less than 3 times upper limit of normal (ULN)
* Bilirubin less than 1.5 times ULN

Renal:

* Creatinine less than 1.5 times ULN OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Fractional shortening at least 29% by echocardiogram OR
* Ejection fraction at least 50% by MUGA
* No prior cardiac dysfunction, even if presently controlled

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No prior anthracycline more than 450 mg/m^2

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent cancer therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-12; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Meyers, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee